CLINICAL TRIAL: NCT03014232
Title: Comparison Cytokine Clearance Between Sustained Low-Efficiency Diafiltration (SLED-f) Using High Cut-off Dialyzer and High-flux Dialyzer in Septic AKI Patients
Brief Title: Comparison Cytokine Clearance Between SLED-f Using High Cut-off Dialyzer and High-flux Dialyzer in Septic AKI Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Khajohn Tiranathanagul, Assistant Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 271/54
Record Dates: First submitted 2017-01-04; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Sepsis; Acute Kidney Injury
Keywords: sustained low-efficiency diafiltration (SLED-f); high cut-off dialyzer; cytokines
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLED-f with HCO dialyzer (Experimental): Online sustained low-efficiency diafiltration (online SLED-f) using novel high cut-off dialyzer which had larger pore size than standard high-flux dialyzer was assigned as the new intervention to compare the efficacy of cytokine removals with the control arm.
  Interventions: Procedure: SLED-f with HCO dialyzer
- SLED-f with HF dialyzer (Active Comparator): Online sustained low-efficiency diafiltration (online SLED-f) using standard high-flux dialyzer in septic acute kidney injury patients was assigned as the control group
  Interventions: Procedure: SLED-f with HF dialyzer

INTERVENTIONS:
Procedure: SLED-f with HCO dialyzer — Online SLED-f with high cut-off dialyzers were performed using the Fresenius 5008S hemodiafiltration machines (Fresenius Medical Care, Bad Homburg, Germany). Super-flux, Sureflux 150FH (Nipro Corporation, Osaka, Japan; cellulose triacetate material, pore size 78 A◦, Kuf 66.9 mL/hr/mmHg, surface area 1.5 m2) were used. Dialysis time and blood flow rate were 6 hours and 200 mL/min, respectively. The predilution reinfusion fluid rate and dialysate flow rate were 80 and 220 mL/min, respectively (the total dialysis fluid flow rate was 300 mL/min).
  Arms: SLED-f with HCO dialyzer
Procedure: SLED-f with HF dialyzer — Online SLED-f with standard high-flux dialyzers were performed using the same Fresenius 5008S hemodiafiltration machines (Fresenius Medical Care, Bad Homburg, Germany). High-flux ELISIO 150H (Nipro Corporation, Osaka, Japan; polynephron material, pore size 50-60 A◦, Kuf 67 mL/hr/mmHg, surface area 1.5 m2) were used. Dialysis time and blood flow rate were 6 hours and 200 mL/min, respectively. The predilution reinfusion fluid rate and dialysate flow rate were 80 and 220 mL/min, respectively (the total dialysis fluid flow rate was 300 mL/min).
  Arms: SLED-f with HF dialyzer

SUMMARY:
Hypercytokinemia contributes a major role in the pathogenesis and is associated with the high mortality in sepsis-related acute kidney injury(AKI). This pilot randomized controlled trial was conducted in sepsis-related AKI patients to compare the efficacy of cytokine removal including interleukin(IL)-6, IL-8, IL-10, and tumor necrotic factor(TNF)-α by six-hour SLED-f between using HCO dialyzer(HCO-SLED-f) and HF dialyzer(HF-SLED-f).

DETAILED DESCRIPTION:
Hypercytokinemia contributes a major role in the pathogenesis and is associated with the high mortality in sepsis-related acute kidney injury(AKI). Reductions of these cytokines have been reported to improve clinical outcomes. Online sustained low-efficiency diafiltration(SLED-f) using traditional high-flux(HF) dialyzer could remove some cytokines. Interestingly, the potential of enhancing cytokine removal by using newly designed high cut-off(HCO) dialyzer that could theoretically remove larger molecular weight solutes has never been studied in SLED-f before.This pilot randomized controlled trial was conducted in sepsis-related AKI patients to compare the efficacy of cytokine removal including interleukin(IL)-6, IL-8, IL-10, and tumor necrotic factor(TNF)-α by six-hour SLED-f between using HCO dialyzer(HCO-SLED-f,n=8) and HF dialyzer(HF-SLED-f,n=8).

ELIGIBILITY:
Inclusion Criteria:

* Sepsis
* Acute kidney injury stage 3

Exclusion Criteria:

* Profound hemodynamic instability with more than one inotropic drug
* Pregnancy
* Breast-feeding
* Delayed receiving antibiotic up to 6 hours after beginning of septic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
IL-6 Clearance | At 30 minutes after the treatment was started
  Simultaneous pre-and post-dialyzer blood samples from arterial and venous sampling ports were collected at 30 minutes after the treatment was started for determination of dialyzer clearances.

SECONDARY OUTCOMES:
Urea percentage of reduction ratio | At time 0-hour and 6-hour of the study SLED-f session
  Blood samples were taken from patients before and at the end of 6-hour in the first online SLED-f session. The percentage of reduction ratio were calculated from the before and ending samples.
Beta2-microglobulin percentage of reduction ratio | At time 0-hour and 6-hour of the study SLED-f session
  Blood samples were taken from patients before and at the end of 6-hour in the first online SLED-f session. The percentage of reduction ratio were calculated from the before and ending samples.
IL-10 Clearances | At 30 minutes after the treatment was started
  Simultaneous pre-and post-dialyzer blood samples from arterial and venous sampling ports were collected at 30 minutes after the treatment was started for determination of dialyzer clearances.
TNF-α Clearances | At 30 minutes after the treatment was started
  Simultaneous pre-and post-dialyzer blood samples from arterial and venous sampling ports were collected at 30 minutes after the treatment was started for determination of dialyzer clearances.
Intradialytic hypotension | During 6 hours of SLED-f session
  The hypotensive events were records
Albumin loss in spent dialysate | During 6 hours of SLED-f session
  Continuous sampling of spent effluent dialysate and ultrafiltrate were carried out with a collection pump inserted into the effluent outlet line via a special connector for total albumin loss determination

CONTACTS AND LOCATIONS:
Overall Officials: Khajohn Tiranathanagul, MD, Principal Investigator — Chulalongkorn University; Jeeraluk Tunpornchai, MD, Principal Investigator — Chulalongkorn University

IPD SHARING:
Plan to Share IPD: No